CLINICAL TRIAL: NCT03152175
Title: Post-traumatic Stress Disorders in Police, Correctional Service Officers, and 911 Operators: A Cost-effectiveness and Efficacy Comparison of Treatment as Usual and a Novel Intervention
Brief Title: Posttraumatic Stress Disorders in Police, Correctional Service Officers, and 911 Operators
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Institut de Recherche Robert-Sauvé en Santé et en Sécurité du Travail (Other)
Responsible Party: Principal Investigator, Alain Brunet, Ph.D., Primary Investigator and Full Professor, Department of Psychiatry, McGill University., Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRPL-007
Record Dates: First submitted 2017-03-30; First posted 2017-05-12 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Trauma and Stressor Related Disorders; Post-traumatic Stress Disorders; Adjustment Disorders; Acute Stress Disorder
Keywords: Memory Reconsolidation; Propranolol; Police officers; 911 operators; Efficacy; Cost-effectiveness
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Stress Disorders, Post-Traumatic; Adjustment Disorders; Stress Disorders, Traumatic, Acute | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Repeated measures parallel design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol Hydrochloride (Experimental): 1mg / kg of propranolol hydrochloride administered as a capsule 60 minutes prior to memory reactivation
  Interventions: Drug: Propranolol Hydrochloride
- Placebo (Placebo Comparator): Placebo manufactured as a capsule to mimic 1mg/kg of propranolol hydrochloride administered 60 minutes prior to memory reactivation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol Hydrochloride — 1mg / kg of propranolol hydrochloride, oral capsule
  Other Names: Teva-propranolol
  Arms: Propranolol Hydrochloride
Drug: Placebo — 1mg / kg of matched placebo, oral capsule
  Arms: Placebo

SUMMARY:
Police officers, correctional service officers, and 911-operators are at increased risk for suffering from trauma-related disorders due to their direct and indirect exposure to life-threatening events, such as shootings, violent assaults, or car accidents, among others. Typical treatments for post-traumatic stress disorders include psychotherapy and pharmacological therapies (i.e., antidepressants). Although these interventions are effective for many sufferers, they all have limitations. Thus, the investigators propose to explore the usefulness of a new therapeutic technique, reconsolidation blockade, which involves reactivating the trauma memory while under the influence of propranolol. Objectives and hypotheses: To explore the efficacy and cost-effectiveness of reconsolidation blockade therapy as an adjunct treatment for trauma- and stressor-related disorders as defined in the Diagnostic and Statistical Manual Mental Disorders-5. The investigators hypothesize that, compared to the control group, 5 weekly trauma-memory reactivations under propranolol treatment will confer a significant reduction in trauma-related symptoms and significantly more health-related economic benefits. Stress symptoms and health-related costs will be assessed at 7, 26 and 52 weeks after study inclusion. In this study, the investigators will also explore the effects of reconsolidation blockade with propranolol on various neuropsychological functions.

ELIGIBILITY:
Inclusion Criteria:

* Understands and reads French
* Currently or previously worked for the Quebec City Police Department, or the 911 dispatch for Quebec City, or another police department or 911 dispatch in the province of Quebec, or for the Quebec Ministry of Public Security as a correctional service officer
* Meets criteria for a trauma-and stressor-related disorder, such as: Acute Stress Disorder, Posttraumatic Stress Disorder, Adjustment Disorder, Other Trauma- and Stressor-Related Disorder, as defined by the Diagnostic and Statistical Manual for Mental Disorders, 5th edition.
* The trauma-and stressor-related disorder must be due to a work-related event.
* A score of at least 4 (moderately ill) on the Clinical Global Impressions-Severity Scale.
* Participants who are currently taking a Selective Serotonin Reuptake Inhibitors or Selective Norepinephrine Reuptake Inhibitors (antidepressants) must accept to skip their morning dose on the days that they receive the study's intervention.

Exclusion Criteria:

* Systolic blood pressure < 100mm Hg (millimeter of mercury) at visit 0.
* Heart rate < 55 bpm (beats per minute) at visit 0.
* Medical conditions that contraindicate propranolol administration, as determined by the treating physician.
* Previous diagnosis of a traumatic brain injury (TBI).
* Previous adverse reaction or non-compliance with a beta-blocker.
* Medications that can have an dangerous interaction with propranolol.
* Fertile women who are not using an adequate contraceptive methods.
* Pregnant women.
* Nursing women.
* The following psychiatric conditions: past or present bipolar disorder, past or present psychotic disorder, present substance abuse or dependence, actively suicidal, past or present neurological disorder, complex posttraumatic stress disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
EuroQol five dimensions questionnaire with five-level scale | The weighted average of the questionnaire responses will be calculated over a 12 month period
  This questionnaire is a standardized instrument for measuring generic health status

SECONDARY OUTCOMES:
Post-traumatic Checklist for the Diagnostic and Statistical Manual for Mental Disorders - 5th edition (PCL-5) | Change from baseline (week 0) to weeks 1, 2, 3, 4 , 5, 7, 26, and 52.
  Measure of trauma and stressor related symptoms
Hopkins Symptom Checklist - 25 (HSCL - 25). | Change from baseline (week 0) to weeks 1, 2, 3, 4 , 5, 7, 26, and 52.
  Measure of depression and anxiety symptom severity
Operational Police Stress Questionnaire (PSQ-OP) | Change from baseline (week 0) to weeks 7, 26, and 52.
  Measure of severity of occupational stress

OTHER OUTCOMES:
Social Functioning Questionnaire (SFQ) | Change from baseline (week 0) to weeks 7, 26, and 52.
  Measure of psycho-social functional
Rey's 15-Item Memory test | Change from baseline (week 0) to weeks 7 and 52.
  Measure of verbal learning and memory
The Logical Memory subtest of the Wechsler Memory Scale - III | Change from baseline (week 0) to weeks 7 and 52.
  Measure of verbal learning and memory
Trail Making Test | Change from baseline (week 0) to weeks 7 and 52.
  Measure of mental flexibility
Color-Word Interference Test of the Delis-Kaplan Executive Function System | Change from baseline (week 0) to weeks 7 and 52.
  Measure of selective attention
Coding subtest of the Wechsler Adult Intelligence Scale-IV | Change from baseline (week 0) to weeks 7 and 52.
  Measure of working memory
Attention subtest of the Paced Auditory Serial Addition Test (PASAT) | Change from baseline (week 0) to weeks 7 and 52.
  Measure of working memory, divided attention, and information processing speed
D2 Test of attention | Change from baseline (week 0) to weeks 7 and 52.
  Measure of selective and sustained attention
Verbal Fluency Test | Change from baseline (week 0) to weeks 7 and 52.
  Measure of verbal ability and executive control
Subjective Units of Distress Scale | Changes from week 1 to weeks 2, 3, 4 and 5.
  Measure of subjective distress from exposure to an event

CONTACTS AND LOCATIONS:
Overall Officials: Alain Brunet, PhD., Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided